CLINICAL TRIAL: NCT02712411
Title: A Randomized, Open-Label, Crossover, Single-Dose Study to Compare Pharmacokinetic Properties and Safety After Administration of HCP1303 Capsule and Co-administration of HGP1201 Tablet, HIP1402 Capsule in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety of HCP1303 and Co-administration of HGP1201, HIP1402 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-TASU-102
Record Dates: First submitted 2016-02-24; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-02

CONDITIONS: Erectile Dysfunction; Prostatic Hyperplasia
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): T → R
  T : HCP1303 R : HGP1201 + HIP1402
  Interventions: Drug: HCP1303; Drug: HGP1201; Drug: HIP1402
- Sequence 2 (Experimental): R → T
  T : HCP1303 R : HGP1201 + HIP1402
  Interventions: Drug: HCP1303; Drug: HGP1201; Drug: HIP1402

INTERVENTIONS:
Drug: HCP1303
Drug: HGP1201
Drug: HIP1402

SUMMARY:
To investigate the pharmacokinetic properties and safety after administration of HCP1303 and co-administration of HGP1201, HIP1402 in healthy male volunteers

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetic properties and safety after administration of HCP1303 and co-administration of HGP1201, HIP1402 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 20~55 years
2. The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
3. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
4. Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. History of relevant drug allergies or clinically significant hypersensitivity reaction.
3. Glomerular filtration rate is under 60ml/min which is calculated by serum creatinine value.
4. Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.
5. SBP: lower than 90mmHg or higher than 150mmHg, DBP: lower thatn 60mmHg or higher than 100mmHg
6. Subjects who judged ineligible by the investigator.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
AUClast | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
Cmax | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose

SECONDARY OUTCOMES:
AUCinf | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
tmax | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
t1/2 | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
Cl/F | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
Vd/F | Pre-dose(0h), 0.5, 1, 1.5, 2, 2.5, 3, 4, 4.5, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Minsu Park, M.D., Ph.D., Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seodaemun-Gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No